CLINICAL TRIAL: NCT03355820
Title: Persistence of Immune Response to GSK Biologicals' HPV Vaccine in Healthy Chinese Female Subjects From the HPV-058 Study
Brief Title: A Follow-up Extension Study to Evaluate the Persistence of Immune Response to GSK Biologicals' HPV Vaccine in Healthy Chinese Female Subjects Who Received Three Doses of the Vaccine in the HPV-058 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 207347; 2017-000255-50 (EudraCT Number)
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Results first posted 2019-06-10 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Immune response; Cervarix; Persistence; Chinese; Human papillomavirus
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV Group (Experimental): Healthy Chinese female subjects, including and above 17 years of age at the time of enrollment, who received all three doses of the Cervarix vaccine in the HPV-058 (NCT00996125) primary study.
  Interventions: Procedure: Blood sampling for antibody determination

INTERVENTIONS:
Procedure: Blood sampling for antibody determination — In order to assess the persistence of immune responses seven to eight years after the last vaccine dose against HPV-16/18, a blood sample (~5 mL) will be taken from all the subjects, at Day 1.

SUMMARY:
The purpose of this study is to evaluate the persistence of immune response in subjects who received the HPV-16/18 vaccine, seven to eight years after the last dose of primary vaccination in the HPV-058 study. No new subjects will be enrolled in this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects/subject's parents/legally acceptable representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject or subject's parents/LAR(s) prior to performing any study specific procedure.
* Written informed assent obtained from the subjects below the legal age of consent.
* Subjects who received all three doses of the HPV-16/18 vaccine in the HPV-058 study.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine which may have an impact on the study objectives) during the period starting 30 days (Day 29 to Day 1) before the study visit.
* Concurrently participating in another clinical study, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Previous vaccination against HPV outside the HPV-058 study.
* Subjects with contraindications related to blood draw such as blood disorders and anticoagulants use.

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Taizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20720

REFERENCES:
- [Background] Hu Y, Zhang X, He Y, Ma Z, Xie Y, Lu X, Xu Y, Zhang Y, Jiang Y, Xiao H, Struyf F, Folschweiller N, Jiang J, Poncelet S, Karkada N, Jastorff A, Borys D. Long-term persistence of immune response to the AS04-adjuvanted HPV-16/18 vaccine in Chinese girls aged 9-17 years: Results from an 8-9-year follow-up phase III open-label study. Asia Pac J Clin Oncol. 2020 Dec;16(6):392-399. doi: 10.1111/ajco.13398. Epub 2020 Aug 11. PMID 32780946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in China.
Pre-assignment Details: 228 subjects were included in the Enrolled Set, 1 subject was excluded from all statistical analyses, thus 227 subjects formed the Exposed Set.
Period: Overall Study
Arm/Group | HPV Group
Started | 227
Completed | 227
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HPV Group
Number analyzed (Participants) | 227
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.6 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 227

OUTCOME MEASURES:

1. Primary Outcome: Number of Seropositive Subjects for Anti-HPV-16 Antibodies at Day 1 in HPV-093 (NCT03355820) Study
Description: A seropositive subject is defined as a subject whose antibody concentration is equal to or above the cut-off value of 19 Enzyme Linked Immunosorbent Assay units per milliliter (EL.U/mL).
Time Frame: At Day 1 in HPV-093 (NCT03355820) study (i.e. 7 to 8 years after completion of the vaccination schedule in HPV-058 [NCT00996125] study)
Population: The analysis was performed on the Per-Protocol Set (PPS) for analysis of immunogenicity, which included all evaluable subjects who were included in the according to protocol (ATP) immunogenicity analysis of the primary vaccination study HPV-058 (NCT00996125), and with serology results available at this blood sampling time point.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Group
Number analyzed (Participants) | 223
Participants | 223

2. Primary Outcome: Number of Seropositive Subjects for Anti-HPV-18 Antibodies at Day 1 in HPV-093 (NCT03355820) Study
Description: A seropositive subject is defined as a subject whose antibody concentration is equal to or above the cut-off value of 18 EL.U/mL.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Group
Number analyzed (Participants) | 223
Participants | 223

3. Primary Outcome: Anti-HPV-16 Antibody Concentrations at Day 1 in HPV-093 (NCT03355820) Study
Description: Anti-HPV-16 antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in EL.U/mL.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV Group
Number analyzed (Participants) | 223
EL.U/mL | 1236.3 [1121.8 to 1362.4]

4. Primary Outcome: Anti-HPV-18 Antibody Concentrations at Day 1 in HPV-093 (NCT03355820) Study
Description: Anti-HPV-18 antibody concentrations are presented as GMCs, expressed in EL.U/mL.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV Group
Number analyzed (Participants) | 223
EL.U/mL | 535.6 [478.6 to 599.4]

5. Secondary Outcome: Number of Seropositive Subjects for Anti-HPV-16 Antibodies at Day 1 in HPV-093 (NCT03355820) and at Year 6 in HPV-039 (NCT00779766) Studies
Description: A seropositive subject is defined as a subject whose antibody concentration is equal to or above the cut-off value of 19 EL.U/mL.
  The number of seropositive subjects at Day 1 in the present study was compared with the number of seropositive subjects from the immunogenicity subset in HPV-039 (NCT00779766) study at Year 6.
  Data corresponding to Day 1 time point of the present study can also be found in the primary outcome measure.
  Data at Year 6 in subjects from the immunogenicity subset in HPV-039 study can be found in the respective NCT record NCT00779766 (please refer to Outcome measure 38, Row "≥19 EL.U/mL, sero-, [Month 72]" and Row "≥19 EL.U/mL, sero+, [Month 72]").
Time Frame: At Day 1 in HPV-093 (NCT03355820) study (i.e. 7 to 8 years after completion of the vaccination schedule in HPV-058 [NCT00996125] study) and at Year 6 in HPV-039 (NCT00779766) study
Population: The analysis was performed on the PPS for analysis of immunogenicity in HPV-093 study and on the ATP cohort for analysis of immunogenicity which included all evaluable subjects in the immunogenicity subset of HPV-039 study. For Year 6 data in HPV-039 study, please refer to the Outcome measure 38 in NCT00779766 record.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Group
Number analyzed (Participants) | 223
Participants | 223

6. Secondary Outcome: Number of Seropositive Subjects for Anti-HPV-18 Antibodies at Day 1 in HPV-093 (NCT03355820) and at Year 6 in HPV-039 (NCT00779766) Studies
Description: A seropositive subject is defined as a subject whose antibody concentration is equal to or above the cut-off value of 18 EL.U/mL.
  The number of seropositive subjects at Day 1 in the present study was compared with the number of seropositive subjects from the immunogenicity subset in HPV-039 (NCT00779766) study at Year 6.
  Data corresponding to Day 1 time point of the present study can also be found in the primary outcome measure.
  Data at Year 6 in subjects from the immunogenicity subset in HPV-039 study can be found in the respective NCT record NCT00779766 (please refer to Outcome measure 39, Row "≥ 18 EL.U/mL, sero- [Month 72]" and Row "≥ 18 EL.U/mL, sero+ [Month 72]).
Time Frame: as for outcome 5
Population: The analysis was performed on the PPS for analysis of immunogenicity in HPV-093 study and on the ATP cohort for analysis of immunogenicity which included all evaluable subjects in the immunogenicity subset of HPV-039 study. For Year 6 data in HPV-039 study, please refer to the Outcome measure 39 in NCT00779766 record.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV Group
Number analyzed (Participants) | 223
Participants | 223

7. Secondary Outcome: Concentration of Antibodies Against HPV-16 at Day 1 in HPV-093 (NCT03355820) and at Year 6 in HPV-039 (NCT00779766) Studies
Description: Anti-HPV-16 antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in EL.U/mL.
  Anti-HPV-16 antibody concentrations at Day 1 in the present study were compared with the anti-HPV-16 antibody concentrations obtained as per the analysis performed on the immunogenicity subset in HPV-039 (NCT00779766) study at Year 6.
  Data corresponding to Day 1 time point of the present study can also be found in the primary outcome measure.
  Data at Year 6 in subjects from the immunogenicity subset in HPV-039 study can be found in the respective NCT record NCT00779766 (please refer to Outcome measure 40, Row "HPV-16, sero-, [Month 72]" and Row "HPV-16, sero+, [Month 72]").
Time Frame: as for outcome 5
Population: The analysis was performed on the PPS for analysis of immunogenicity in HPV-093 study and on the ATP cohort for analysis of immunogenicity which included all evaluable subjects in the immunogenicity subset of HPV-039 study. For Year 6 data in HPV-039 study, please refer to the Outcome measure 40 in NCT00779766 record.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV Group
Number analyzed (Participants) | 223
EL.U/mL | 1236.3 [1121.8 to 1362.4]

8. Secondary Outcome: Concentration of Antibodies Against HPV-18 at Day 1 in HPV-093 (NCT03355820) and at Year 6 in HPV-039 (NCT00779766) Studies
Description: Anti-HPV-18 antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in EL.U/mL.
  Anti-HPV-18 antibody concentrations at Day 1 in the present study were compared with the anti-HPV-18 antibody concentrations obtained as per the analysis performed on the immunogenicity subset in HPV-039 (NCT00779766) study at Year 6.
  Data corresponding to Day 1 time point of the present study can also be found in the primary outcome measure.
  Data at Year 6 in subjects from the immunogenicity subset in HPV-039 study can be found in the respective NCT record NCT00779766 (please refer to Outcome measure 40, Row "HPV-18, sero-, [Month 72]" and Row "HPV-18, sero+, [Month 72]").
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV Group
Number analyzed (Participants) | 223
EL.U/mL | 535.6 [478.6 to 599.4]

ADVERSE EVENTS:
Time Frame: At Day 1
Description: There were no adverse events (AEs) data collected during the entire study period (i.e. at Day 1).
  Only SAEs related to study procedures or concomitant GSK medications/vaccines and events with a fatal outcome were recorded and collected during the entire study period (i.e. at Day 1).
Arm/Group | HPV Group
All-Cause Mortality (participants affected / at risk) | 0/227
Serious Adverse Events (participants affected / at risk) | 0/227
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT03355820/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT03355820/SAP_001.pdf